CLINICAL TRIAL: NCT01510626
Title: Omalizumab With Oral Food Immunotherapy With Food Allergies Open Label Safety Study in a Single Center
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kari Christine Nadeau, Associate Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22872; NCT02062814 (obsolete NCT alias)
Record Dates: First submitted 2011-11-29; First posted 2012-01-16 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Immune System Diseases
Keywords: Multiple food allergies
MeSH Terms: conditions — Immune System Diseases | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- One (Experimental)
  Interventions: Dietary Supplement: Food proteins; Drug: Omalizumab

INTERVENTIONS:
Dietary Supplement: Food proteins — Food proteins
Drug: Omalizumab — Drug

SUMMARY:
The long-term goal of the investigators study is to develop a better and safer treatment for, and to potentially cure patients with single or multiple food allergies. The investigators hypothesize that the application of this protocol will allow patients with severe and single or multiple food allergies to be safely and rapidly desensitized.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe peanut and/or egg and/or milk and/or tree nut and/or seed allergic subjects between the ages of 4 to 55 years old.
* Sensitivity to food allergen will be documented by a positive skin prick test result or allergen-specific ImmunoCAP IgE level, with 7 kU/L as a lower limit of eligibility.

Exclusion Criteria:

* No absolute contraindications are known. However, the risk of serious systemic anaphylactic reactions to food allergens suggests a number of preexisting conditions that should be considered relative contraindications. Among those conditions are acute infections, autoimmune disease, severe cardiac disease, and treatment with beta-adrenergic antagonistic drugs (beta-blockers).
* Subjects with a total IgE at screening of >2,000 kU/L
* Previous reaction to omalizumab
* Subjects having a history of severe anaphylaxis to food allergens that will be desensitized in this study requiring intubation or admission to an ICU, frequent allergic or non-allergic urticaria, or history consistent with poorly controlled persistent asthma.

Ages: 4 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2011-11; Primary Completion 2014-04 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of adverse events in the treatment population | 2 years

SECONDARY OUTCOMES:
Number of subjects who reach 2g or more of food flour | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Andorf S, Manohar M, Dominguez T, Block W, Tupa D, Kshirsagar RA, Sampath V, Chinthrajah RS, Nadeau KC. Observational long-term follow-up study of rapid food oral immunotherapy with omalizumab. Allergy Asthma Clin Immunol. 2017 Dec 21;13:51. doi: 10.1186/s13223-017-0223-8. eCollection 2017. PMID 29296107